CLINICAL TRIAL: NCT00399061
Title: Efficacy of Optive Versus Systane Concomitant With Restasis (Cyclosporine A) for the Treatment of Dry Eye Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Robert Schultze, MD, Slingerlands Medical Building
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5278
Record Dates: First submitted 2006-11-09; First posted 2006-11-14 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Active Comparator): Systane
  Interventions: Drug: Systane, Optive, Restasis
- 2 (Active Comparator): Optive
  Interventions: Drug: Systane, Optive, Restasis
- 3 (Placebo Comparator): Restasis
  Interventions: Drug: Systane, Optive, Restasis

INTERVENTIONS:
Drug: Systane, Optive, Restasis — Systane 30ml (in the eye) instill one drop twice a day in morning and evening Optive 15ml (in the eye) instill one drop twice a day in morning and evening Restasis 0.4ml (in the eye) instill one drop twice a day in morning and evening more frequently if needed

SUMMARY:
The purpose of this study is to evaluate the efficacy of Optive versus Systane used concomitantly with topical cyclosporine for the treatment of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* · Males or females > 18 years old

  * Score of at least 2 and no more than 4 on the SESOD at the initial screening visit (mild to severe patients)
  * At least Grade 2 conjunctival staining
  * Likely to complete all study visits and able to provide informed consent

Exclusion Criteria:

* · Prior unsuccessful use of topical cyclosporine (defined as patients taking it at least 3 months and saw no improvements)

  * Current use of topical cyclosporine
  * Known contraindications to any study medication or ingredients
  * Female of child bearing potential not using reliable methods of birth control, or pregnant or lactating females.
  * Planned use of contact lenses (unless discontinued use ³ 30 days prior to randomization)
  * Active ocular diseases or uncontrolled systemic disease (blepharitis patients that are actively being treated or disease that is uncontrollable)
  * Ocular surgery within the past 3 months,
  * Active ocular allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Efficacy | 1 yr 3 months

SECONDARY OUTCOMES:
Dry eye symptoms | 1yr 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schultze, MD, Principal Investigator — Slingerlands Medical Building
Locations (1):
- Dr. Schultze, Slingerlands, New York, United States